CLINICAL TRIAL: NCT06718998
Title: Evaluation of Different Dose Escalation Regimens for NNC0519-0130 in Participants With Overweight and Obesity
Brief Title: A Research Study Comparing Different Ways of Increasing the Dose of NNC0519-0130 in Participants With Overweight or Obesity
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9541-7760; U1111-1298-9340 (Other: World Health Organization (WHO)); 2023-508940-23 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1: NNC0519-0130 (Experimental): Participants will receive once-weekly subcutaneous (s.c) injections of NNC0519-0130 following a predetermined dose escalation regimen 1 in the main and extension phase.
  Interventions: Drug: NNC0519-0130
- Arm 2: NNC0519-0130 (Experimental): Participants will receive once-weekly s.c injections of NNC0519-0130 following a predetermined dose escalation regimen 2 in the main phase and extension phase.
  Interventions: Drug: NNC0519-0130
- Arm 3: NNC0519-0130 (Experimental): Participants will receive twice-weekly s.c injections of NNC0519-0130 following a predetermined dose escalation regimen 3 in the main phase and extension phase.
  Interventions: Drug: NNC0519-0130
- Arm 4: NNC0519-0130 (Experimental): Participants will receive once-weekly s.c injections of NNC0519-0130 following a predetermined dose escalation regimen 4 in the main and extension phase.
  Interventions: Drug: NNC0519-0130

INTERVENTIONS:
Drug: NNC0519-0130 — Participants will receive once-weekly or twice weekly NNC0519-0130 subcutaneously.

SUMMARY:
Novo Nordisk is developing a new study medicine NNC0519-0130 to improve the treatment options for people living with type 2 diabetes and people with excess body weight. This study will look at the safety and tolerability of NNC0519-0130. The purpose of this study is to investigate if different ways of increasing the dose of NNC0519-0130 in the main and extension phase can lessen the side effects that may occur when people take NNC0519-0130. There will be four different ways of increasing the dose of the study medicine and participants will get assigned to one of these - which one the participants get is decided by chance. This study will last for about 24 weeks.

ELIGIBILITY:
Inclusion criteria:

* Female of non-childbearing potential, or male.
* Age 18-64 years (both inclusive) at the time of signing the informed consent.
* Body mass index (BMI) between 27.0 and 44.9 kilogram per square meter (kg/m^2) (both inclusive) at screening. Overweight should be due to excess adipose tissue, as judged by the investigator.
* Considered to be otherwise healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion criteria:

* Any disorder, unwillingness or inability which in the investigator's opinion, might jeopardise the participant's safety or compliance with the protocol.
* Glycated haemoglobin (HbA1c) greater than or equal to (>=) 6.5 percentage (48 millimoles per mole [mmol/mol]) at screening.
* Use of prescription medicinal products or non-prescription drugs, except routine vitamins, occasional use of paracetamol, NSAIDs (nonsteroidal anti-inflammatory drugs), acetylsalicylic acid, or topical medication not reaching systemic circulation, within 14 days before screening.
* Presence or history of any clinically relevant respiratory, metabolic, renal, hepatic, cardiovascular, gastrointestinal, or endocrinological conditions.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2026-01-08 (Estimated); Study Completion 2026-01-08 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events (AEs) | From randomisation (week 0) to week 18
  Measured as number of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com